CLINICAL TRIAL: NCT01642004
Title: An Open-Label Randomized Phase III Trial of BMS-936558 (Nivolumab) Versus Docetaxel in Previously Treated Advanced or Metastatic Squamous Cell Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of BMS-936558 (Nivolumab) Compared to Docetaxel in Previously Treated Advanced or Metastatic Squamous Cell Non-small Cell Lung Cancer (NSCLC) (CheckMate 017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-017; 2011-004792-36 (EudraCT Number)
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously (IV) every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends. Eligible patients may receive nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Biological: Nivolumab
- Arm B: Docetaxel (Experimental): Docetaxel 75 mg/m^2 concentrate for solution for intravenous infusion every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends. Eligible patients may receive nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558
  Arms: Arm A: Nivolumab
Drug: Docetaxel
  Other Names: Taxotere®
  Arms: Arm B: Docetaxel

SUMMARY:
The purpose of the study is to compare the overall survival of BMS-936558 as compared with Docetaxel in subjects with squamous cell non-small cell lung cancer (NSCLC), after failure of prior platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Subjects with histologically or cytologically-documented squamous cell NSCLC who present with Stage IIIB/IV disease or with recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection or definitive chemoradiation therapy for locally advanced disease)
* Disease recurrence or progression during/after one prior platinum doublet-based chemotherapy regimen for advanced or metastatic disease
* Measurable disease by computed tomography (CT)/Magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* A formalin fixed, paraffin-embedded (FFPE) tumor tissue block or unstained slides of tumor sample (archival or recent) must be available for biomarker evaluation. Specimens must be received by the central lab prior to randomization. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient

Exclusion Criteria:

* Subjects with untreated central nervous system (CNS) metastases are excluded. Subjects are eligible if CNS metastases are treated and subjects are neurologically returned to baseline for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent)
* Subjects with carcinomatous meningitis
* Subjects with active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of randomization
* Prior therapy with anti-Programmed death-1 (PD-1), anti-Programmed cell death ligand 1 (PD-L1), anti-Programmed cell death ligand 2 (PD-L2), anti-CD137, or anti-Cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Prior treatment on the first line study CA184104 first line NSCLC study
* Prior treatment with Docetaxel
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Treatment with any investigational agent within 14 days of first administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (39):
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - City Of Hope, Duarte, California
  - Local Institution - 0020, Duarte, California
  - Local Institution - 0009, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0004, Tampa, Florida
  - Local Institution - 0153, Marietta, Georgia
  - Local Institution - 0100, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Local Institution - 0003, Baltimore, Maryland
  - Local Institution - 0036, Boston, Massachusetts
  - Local Institution - 0084, Boston, Massachusetts
  - Local Institution - 0150, Boston, Massachusetts
  - Local Institution - 0016, Mineola, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Local Institution - 0006, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Local Institution - 0008, Durham, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0011, Philadelphia, Pennsylvania
  - Guthrie Medical Group, Pc, Sayre, Pennsylvania
  - Local Institution - 0082, Columbia, South Carolina
  - Local Institution - 0087, Chattanooga, Tennessee
  - Local Institution - 0005, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Local Institution - 0032, Nashville, Tennessee
  - Local Institution - 0012, Dallas, Texas
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0086, Houston, Texas
  - Local Institution - 0017, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Local Institution - 0001, Seattle, Washington
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Local Institution - 0033, Morgantown, West Virginia
- Argentina (5):
  - Local Institution - 0116, Capital Federal, Buenos Aires
  - Local Institution - 0072, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Local Institution - 0164, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0071, Buenos Aires
  - Local Institution - 0141, Córdoba
- Australia (5):
  - Local Institution - 0073, Wollongong, New South Wales
  - Local Institution - 0159, Adelaide, South Australia
  - Local Institution - 0140, Elizabeth Vale, South Australia
  - Local Institution - 0158, Kurralta Park, South Australia
  - Local Institution - 0085, Clayton, Victoria
- Austria (4):
  - Local Institution - 0102, Linz
  - Local Institution - 0104, Salzburg
  - Local Institution - 0049, Vienna
  - Local Institution - 0103, Wels
- Canada (3):
  - Local Institution - 0146, Winnipeg, Manitoba
  - Local Institution - 0147, Montreal, Quebec
  - Local Institution - 0152, Rimouski, Quebec
- Chile (5):
  - Local Institution - 0110, Viña del Mar, Región de Valparaíso
  - Local Institution - 0117, Santiago, Santiago Metropolitan
  - Local Institution - 0131, Santiago, Santiago Metropolitan
  - Local Institution - 0161, Antofagasta
  - Local Institution - 0154, Santiago
- Local Institution - 0111, Prague, Czechia
- France (14):
  - Local Institution - 0053, Avignon Cedes 9
  - Local Institution - 0156, Caen
  - Local Institution - 0025, Dijon
  - Local Institution, Dijon
  - Local Institution - 0093, La Roche-sur-Yon
  - Local Institution - 0022, Lyon
  - Local Institution, Lyon
  - Local Institution - 0023, Marseille
  - Local Institution, Marseille
  - Local Institution - 0160, Pierre-Bénite
  - Local Institution - 0027, Rennes
  - Local Institution, Rennes
  - Local Institution - 0157, Strasbourg
  - Local Institution - 0040, Toulouse
- Germany (7):
  - Local Institution - 0064, Bad Berka
  - Local Institution - 0063, Cologne
  - Local Institution - 0105, Essen
  - Local Institution - 0109, Gerlingen
  - Local Institution - 0048, Großhansdorf
  - Local Institution - 0065, Heidelberg
  - Local Institution - 0162, Krefeld
- Hungary (2):
  - Local Institution - 0095, Budapest
  - Local Institution - 0096, Budapest
- Ireland (2):
  - Local Institution - 0035, Dublin, Dublin
  - Local Institution - 0039, Dublin, Dublin
- Italy (7):
  - Local Institution - 0058, Bologna
  - Local Institution - 0088, Meldola (fc)
  - Local Institution - 0057, Milan
  - Local Institution - 0056, Padua
  - Local Institution - 0055, Perugia
  - Local Institution - 0089, Ravenna
  - Local Institution - 0054, Siena
- Mexico (4):
  - Local Institution - 0106, Leon, Guanajato, Guanajuato
  - Local Institution - 0107, Mexico City, Mexico City
  - Local Institution - 0108, Mexico City, Mexico City
  - Local Institution - 0139, Hermosillo, Sonora
- Netherlands (2):
  - Local Institution - 0052, Amsterdam
  - Local Institution - 0051, Rotterdam
- Local Institution - 0143, Oslo, Norway
- Peru (2):
  - Local Institution - 0099, Arequipa
  - Local Institution - 0061, Lima
- Poland (5):
  - Local Institution - 0126, Gdansk
  - Local Institution - 0130, Krakow
  - Local Institution - 0129, Olsztyn
  - Local Institution - 0124, Szczecin
  - Local Institution - 0127, Warsaw
- Romania (6):
  - Local Institution - 0136, Bucharest
  - Local Institution - 0145, Cluj-Napoca
  - Local Institution - 0138, Constanța
  - Local Institution - 0121, Craiova
  - Local Institution - 0119, Iași
  - Local Institution - 0120, Timișoara
- Russia (4):
  - Local Institution - 0132, Moscow
  - Local Institution - 0133, Moscow
  - Local Institution - 0144, Moscow
  - Local Institution - 0135, Saint Petersburg
- Spain (5):
  - Local Institution - 0044, Barakaldo, Vizcaya
  - Local Institution - 0042, Barcelona
  - Local Institution - 0046, Madrid
  - Local Institution - 0045, Madrid
  - Local Institution - 0041, Seville
- United Kingdom (4):
  - Local Institution - 0047, Cottingham, East Yorkshire
  - Local Institution - 0034, Southampton, Hampshire
  - Local Institution - 0163, Withington, Manchester
  - Local Institution - 0037, Sheffield, Yorkshire

REFERENCES:
- [Derived] Hu S, Tang Z, Harrison JP, Hertel N, Penrod JR, May JR, Juarez-Garcia A, Holdgate O. Economic Evaluation of Nivolumab Versus Docetaxel for the Treatment of Advanced Squamous and Non-squamous Non-small Cell Lung Cancer After Prior Chemotherapy in China. Pharmacoecon Open. 2023 Mar;7(2):273-284. doi: 10.1007/s41669-022-00383-x. Epub 2023 Mar 10. PMID 36897427
- [Derived] Borghaei H, Gettinger S, Vokes EE, Chow LQM, Burgio MA, de Castro Carpeno J, Pluzanski A, Arrieta O, Frontera OA, Chiari R, Butts C, Wojcik-Tomaszewska J, Coudert B, Garassino MC, Ready N, Felip E, Garcia MA, Waterhouse D, Domine M, Barlesi F, Antonia S, Wohlleber M, Gerber DE, Czyzewicz G, Spigel DR, Crino L, Eberhardt WEE, Li A, Marimuthu S, Brahmer J. Five-Year Outcomes From the Randomized, Phase III Trials CheckMate 017 and 057: Nivolumab Versus Docetaxel in Previously Treated Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Mar 1;39(7):723-733. doi: 10.1200/JCO.20.01605. Epub 2021 Jan 15. PMID 33449799
- [Derived] Dercle L, Fronheiser M, Lu L, Du S, Hayes W, Leung DK, Roy A, Wilkerson J, Guo P, Fojo AT, Schwartz LH, Zhao B. Identification of Non-Small Cell Lung Cancer Sensitive to Systemic Cancer Therapies Using Radiomics. Clin Cancer Res. 2020 May 1;26(9):2151-2162. doi: 10.1158/1078-0432.CCR-19-2942. Epub 2020 Mar 20. PMID 32198149
- [Derived] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Derived] Vokes EE, Ready N, Felip E, Horn L, Burgio MA, Antonia SJ, Aren Frontera O, Gettinger S, Holgado E, Spigel D, Waterhouse D, Domine M, Garassino M, Chow LQM, Blumenschein G Jr, Barlesi F, Coudert B, Gainor J, Arrieta O, Brahmer J, Butts C, Steins M, Geese WJ, Li A, Healey D, Crino L. Nivolumab versus docetaxel in previously treated advanced non-small-cell lung cancer (CheckMate 017 and CheckMate 057): 3-year update and outcomes in patients with liver metastases. Ann Oncol. 2018 Apr 1;29(4):959-965. doi: 10.1093/annonc/mdy041. PMID 29408986
- [Derived] Horn L, Spigel DR, Vokes EE, Holgado E, Ready N, Steins M, Poddubskaya E, Borghaei H, Felip E, Paz-Ares L, Pluzanski A, Reckamp KL, Burgio MA, Kohlhaeufl M, Waterhouse D, Barlesi F, Antonia S, Arrieta O, Fayette J, Crino L, Rizvi N, Reck M, Hellmann MD, Geese WJ, Li A, Blackwood-Chirchir A, Healey D, Brahmer J, Eberhardt WEE. Nivolumab Versus Docetaxel in Previously Treated Patients With Advanced Non-Small-Cell Lung Cancer: Two-Year Outcomes From Two Randomized, Open-Label, Phase III Trials (CheckMate 017 and CheckMate 057). J Clin Oncol. 2017 Dec 10;35(35):3924-3933. doi: 10.1200/JCO.2017.74.3062. Epub 2017 Oct 12. PMID 29023213
- [Derived] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: Nivolumab 3 mg/kg solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends. Eligible patients may receive nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
- Docetaxel: Docetaxel 75mg/m^2 solution intravenously every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or study ends.
Period: Randomization
Arm/Group | Nivolumab | Docetaxel
Started (Started=Randomized) | 135 | 137
Completed (Completed= participants that received treatment) | 131 | 129
Not Completed | 4 | 8
Not completed — Adverse Event unrelated to study drug | 1 | 0
Not completed — Participant withdrew consent | 1 | 6
Not completed — No longer meets study criteria | 2 | 2
Period: Treatment
Arm/Group | Nivolumab | Docetaxel
Started | 131 | 129
Participants Transitioned to Nivolumab | 0 | 6
Completed (Completed = continue in the treatment period) | 0 | 0
Not Completed | 131 | 129
Not completed — Disease progression | 95 | 79
Not completed — Study drug toxicity | 10 | 13
Not completed — Death | 1 | 1
Not completed — Adverse event unrelated to study drug | 9 | 13
Not completed — Maximum clinical benefit | 1 | 9
Not completed — Poor/non-compliance | 1 | 0
Not completed — No longer meets study criteria | 1 | 2
Not completed — Other reasons | 2 | 0
Not completed — Not reported | 0 | 3
Not completed — Participant request to discontinue study treatment | 6 | 4
Not completed — Participant withdrew consent | 5 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Docetaxel | Total
Number analyzed (Participants) | 135 | 137 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.33) | 64.4 (8.28) | 63.3 (8.36)
Age, Customized [Number; unit: Participants]
  <= 18 years | 0 | 0 | 0
  < 65 years | 79 | 73 | 152
  >= 65 AND < 75 years | 45 | 46 | 91
  >= 75 AND < 85 years | 10 | 18 | 28
  >= 85 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 40 | 64
  Male | 111 | 97 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 61 | 60 | 121
  Unknown or Not Reported | 67 | 72 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 122 | 130 | 252
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time in Months for All Randomized Participants at Primary Endpoint
Description: OS was defined as the time between the date of randomization and the date of death from any cause. Participants were censored at the date they were last known to be alive. Median OS time was calculated using Kaplan-Meier (KM) method. Hazard ratio (HR) and the corresponding Confidence Interval (CI) were estimated in a stratified Cox proportional hazards model for distribution of OS in each randomized arm. Interim analysis (Primary Endpoint) was planned to occur after at least 196 deaths, with the actual analysis occurring at 199 deaths.
Time Frame: Randomization until 199 deaths, up to November 2014, approximately 25 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
months | 9.23 [7.33 to 13.27] | 6.01 [5.13 to 7.33]
Statistical Analysis 1: Comparison: Nivolumab vs Docetaxel; Test type: Superiority or Other; p = 0.0002, Log Rank — Stratified by region (US/Canada, Rest Of World (ROW), Europe) and prior treatment regimen (Paclitaxel, Another agent) as entered in the Interactive Voice Response System (IVRS); Hazard Ratio (HR) = 0.59, 96.85% CI 2-sided [0.43 to 0.81] — Stratified Cox proportional hazard model. HR = Nivolumab over Docetaxel

2. Primary Outcome: Overall Survival (OS) Rate in All Randomized Participants
Description: The overall survival rate is the probability that a participant will be alive at 6, 12, and 18 months following randomization. Overall survival was defined as the time between the date of randomization and the date of death as a result of any cause. Survival rates were determined via Kaplan-Meier estimates.
Time Frame: Randomization to 18 months post-randomization, up to June 2015
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent probability of OS
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Percent probability of OS
  6 months | 63.7 [55.0 to 71.2] | 50.7 [42.1 to 58.8]
  12 months | 42.2 [33.8 to 50.4] | 24.3 [17.4 to 31.7]
  18 months | 28.1 [20.8 to 35.8] | 12.5 [7.6 to 18.7]

3. Primary Outcome: Number of Deaths From Any Cause in All Randomized Participants at Primary Endpoint
Description: The number of participants who died from any cause was reported for each arm. Interim analysis (Primary Endpoint) was planned to occur after at least 196 deaths, with the actual analysis occurring at 199 deaths.
Time Frame: Randomization until 199 deaths, up to November 2014, approximately 25 months
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Participants | 86 | 113

4. Secondary Outcome: Objective Response Rate (ORR) in All Randomized Participants
Description: ORR was defined as the percentage of all randomized participants whose Best Overall Response (BOR) was a confirmed Complete Response (CR) or Partial Response (PR). BOR was defined as the best investigator-assessed response designation, recorded between the date of randomization and the date of objectively documented progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or the date of subsequent anti-cancer therapy (excluding on-treatment palliative radiotherapy of non-target bone lesions or Central Nervous System (CNS) lesions), whichever occurred first. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. CIs were computed using the Clopper and Pearson method.
Time Frame: From the date of randomization up to the date of objectively documented progression, up to approximately 103 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Percentage of participants | 20.0 [13.6 to 27.7] | 8.8 [4.6 to 14.8]

5. Secondary Outcome: Time To Response (TTR) in Months for All Confirmed Responders
Description: Time to Response (TTR) for participants demonstrating a response (either CR or PR) was defined as the time from the date of randomization to the date of the first confirmed response. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters.
Time Frame: From the date of randomization to the date of the first confirmed response, up to approximately 12 months
Population: All confirmed responders (participants demonstrating CR or PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 27 | 12
Months | 2.23 [1.6 to 11.8] | 2.09 [1.8 to 9.5]

6. Secondary Outcome: Duration of Objective Response (DOR) in Months for All Confirmed Responders
Description: DOR was defined as the time from the date of first confirmed response to the date of the first documented tumor progression (per RECIST v1.1), as determined by the investigator, or death due to any cause, whichever occurred first. DOR was evaluated only for confirmed responders (i.e. participants with confirmed CR or PR). CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. Participants who neither progressed nor died were censored on the date of their last evaluable tumor assessment.
Time Frame: From the date of first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurred first, up to approximately 94 months
Population: All confirmed responders (participants demonstrating CR or PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 27 | 12
Months | 24.51 [9.76 to 69.65] | 8.41 [3.58 to 14.03]

7. Secondary Outcome: Progression Free Survival Rate (PFSR)
Description: PFSR was defined as the percentage of participants who did not experience disease progression or death from any cause at a given time point following randomization. Progression was assessed by investigators according to RECIST v1.1. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who started any subsequent anti-cancer therapy (including on-treatment palliative radiation therapy (RT) of non-target bone lesions or CNS lesions) without a prior reported progression were to be censored at the last evaluable tumor assessment prior to or on initiation of the subsequent anti-cancer therapy.
Time Frame: From randomization to specified timepoints, up to 84 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Percentage of participants
  6 months | 38.4 [30.0 to 46.8] | 22.6 [15.7 to 30.2]
  12 months | 21.0 [14.3 to 28.6] | 7.2 [3.4 to 12.8]
  18 months | 15.87 [9.9 to 22.8] | 1.8 [0.4 to 5.7]
  24 months | 14.8 [9.1 to 21.8] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.
  36 months | 11.0 [6.1 to 17.5] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.
  48 months | 8.9 [4.5 to 15.1] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.
  60 months | 8.9 [4.5 to 15.1] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.
  72 months | 7.6 [3.5 to 13.7] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.
  84 months | 6.1 [2.4 to 12.2] | NA [NA to NA] — Median, lower and upper limit not reached due to insufficient number of events.

8. Secondary Outcome: Progression-Free Survival (PFS) Time in Months for All Randomized Participants
Description: PFS was defined as the time from the date of randomization to the date of the first documented tumor progression as determined by the investigator per RECIST v1.1 criteria, or death due to any cause. Participants underwent radiographic tumor assessments every 6 weeks (+/- 5 days) from week 9 (+/- 5 days) for the first year on treatment, then every 12 weeks after the first year on treatment until documented disease progression. The PFS curves were estimated using KM method. Two-sided 95% CI for median PFS were computed by Brookmeyer and Crowley method (using log-log transformation). Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who started any subsequent anti-cancer therapy (including on-treatment palliative RT of non-target bone lesions or CNS lesions) without a prior reported progression were to be censored at the last evaluable tumor assessment prior to or on initiation of the subsequent anti-cancer therapy.
Time Frame: From randomization up to the first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurred first, up to approximately 103 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Months | 3.48 [2.14 to 5.06] | 2.83 [2.10 to 3.52]

9. Secondary Outcome: Percentage of Participants Experiencing Disease-related Symptom Improvement by Week 12
Description: Disease-related symptom improvement rate by Week 12 was defined as the percentage of randomized participants who had a 10 point or greater decrease from baseline in average symptom burden index score at any time between randomization and Week 12. The participant portion of the Lung Cancer Symptom Scale (LCSS) consisted of 6 symptom-specific questions that addressed cough, dyspnea, fatigue, pain, hemoptysis, and anorexia, plus 3 summary items on symptom distress, interference with activity level, and global health-related Quality of Life (QoL). The scores range from 0 to 100, with 0 representing the best possible score and 100 being the worst possible score. The average symptom burden index score at each assessment was defined as the mean of the 6 symptom-specific questions of the LCSS. 95% CIs were computed using Clopper-Pearson Method.
Time Frame: From randomization up to Week 12
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
percentage of participants | 18.5 [12.4 to 26.1] | 21.2 [14.7 to 29.0]

10. Secondary Outcome: Overall Survival (OS) Time in Months by Baseline PD-L1 Expression for All Randomized Participants
Description: OS was measured in months for all randomized participants grouped by their baseline PD-L1 expression level. PD-L1 expression was defined as the percent of disease tumor cells demonstrating plasma membrane PD-L1 staining of any intensity using an immunohistochemistry (IHC) assay. OS was defined as the time between the date of randomization and the date of death from any cause. Participants were censored at the date they were last known to be alive. Median OS time was calculated using Kaplan-Meier (KM) method.
Time Frame: From the date of randomization to the date of death from any cause, up to approximately 103 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Months
  PD-L1 expression >= 5%: number analyzed (Participants) | 42 | 39
  PD-L1 expression >= 5% | 9.95 [5.82 to 16.69] | 6.37 [4.50 to 9.03]
  PD-L1 expression < 5%: number analyzed (Participants) | 75 | 69
  PD-L1 expression < 5% | 8.54 [5.49 to 12.62] | 6.14 [5.13 to 8.28]
  PD-L1 not quantifiable at baseline: number analyzed (Participants) | 18 | 29
  PD-L1 not quantifiable at baseline | 9.41 [7.10 to 25.20] | 5.06 [3.02 to 6.11]

11. Secondary Outcome: Objective Response Rate (ORR) by Baseline PD-L1 Expression for All Randomized Participants
Description: ORR was reported for all randomized participants grouped by their baseline PD-L1 expression level. ORR was defined as the percentage of all randomized participants whose Best Overall Response (BOR) was a confirmed Complete Response (CR) or Partial Response (PR). PD-L1 expression in participants was defined as the percent of disease tumor cells demonstrating plasma membrane PD-L1 staining of any intensity using an immunohistochemistry (IHC) assay. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. CIs were computed using the Clopper and Pearson method.
Time Frame: From the date of randomization up to the date of objectively documented progression, up to approximately 103 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Percentage of participants
  PD-L1 expression >= 5%: number analyzed (Participants) | 42 | 39
  PD-L1 expression >= 5% | 21.4 [10.3 to 36.8] | 7.7 [1.6 to 20.9]
  PD-L1 expression < 5%: number analyzed (Participants) | 75 | 69
  PD-L1 expression < 5% | 14.7 [7.6 to 24.7] | 11.6 [5.1 to 21.6]
  PD-L1 not quantifiable at baseline: number analyzed (Participants) | 18 | 29
  PD-L1 not quantifiable at baseline | 38.9 [17.3 to 64.3] | 3.4 [0.1 to 17.8]

12. Secondary Outcome: Progression Free Survival (PFS) Time in Months by Baseline PD-L1 Expression for All Randomized Participants
Description: PFS time was measured for all randomized participants grouped by their baseline PD-L1 expression levels. PFS was defined as the time from the date of randomization to the date of the first documented tumor progression as determined by the investigator per RECIST v1.1 criteria, or death due to any cause. The PFS curves were estimated using KM method. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment. Participants who started subsequent anti-cancer therapy (including on-treatment palliative radiotherapy of non-target bone lesions or CNS lesions) without a prior reported progression were censored at the last evaluable tumor assessment prior to subsequent anti-cancer therapy.
Time Frame: From the date of first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurred first, up to approximately 103 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Months
  PD-L1 expression >= 5%: number analyzed (Participants) | 42 | 39
  PD-L1 expression >= 5% | 5.06 [2.10 to 7.56] | 3.06 [1.94 to 4.63]
  PD-L1 expression < 5%: number analyzed (Participants) | 75 | 69
  PD-L1 expression < 5% | 2.23 [1.94 to 4.73] | 2.92 [2.07 to 3.58]
  PD-L1 not quantifiable at baseline: number analyzed (Participants) | 18 | 29
  PD-L1 not quantifiable at baseline | 5.39 [2.10 to 10.45] | 2.23 [2.04 to 4.40]

13. Post Hoc Outcome: Overall Survival (OS) Time in Months for All Randomized Participants - Extended Collection
Description: OS was defined as the time between the date of randomization and the date of death from any cause. Participants were censored at the date they were last known to be alive. Median OS time was calculated using Kaplan-Meier (KM) method. Hazard ratio (HR) and the corresponding Confidence Interval (CI) were estimated in a stratified Cox proportional hazards model for distribution of OS in each randomized arm. Survival follow-up analysis occurred at the end of the study.
Time Frame: as for outcome 12
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Months | 9.23 [7.33 to 12.62] | 6.01 [5.13 to 7.33]

14. Post Hoc Outcome: Overall Survival (OS) Rate in All Randomized Participants - Extended Collection
Description: The overall survival rate is the probability that a participant will be alive at the specified timepoints following randomization. Overall survival was defined as the time between the date of randomization and the date of death as a result of any cause. Survival rates were determined via Kaplan-Meier estimates.
Time Frame: From the date of randomization up to the specified timepoints, up to 84 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent probability of OS
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 135 | 137
Percent probability of OS
  6 months | 63.7 [55.0 to 71.2] | 50.4 [41.7 to 58.4]
  12 months | 42.2 [33.8 to 50.4] | 24.1 [17.3 to 31.5]
  18 months | 28.1 [20.8 to 35.9] | 12.4 [7.6 to 18.5]
  24 months | 23.0 [16.3 to 30.3] | 8.0 [4.3 to 13.3]
  36 months | 15.6 [10.0 to 22.2] | 5.8 [2.7 to 10.6]
  48 months | 13.1 [8.1 to 19.5] | 4.4 [1.8 to 8.8]
  60 months | 12.3 [7.4 to 18.5] | 3.6 [1.4 to 7.8]
  72 months | 11.4 [6.7 to 17.5] | 2.7 [0.8 to 6.7]
  84 months | 9.6 [5.3 to 15.5] | 0.0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their enrollment to study completion, (up to approximately 103 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 94 months).
Description: All-Cause Mortality = all randomized participants. Serious Adverse Events and Other Adverse Events = all treated participants.
  ARM 1: AEs that occurred on 3mg/kg Nivolumab, ARM 2: AEs that occurred on 480 mg Nivolumab, ARM 3: AEs that occurred on Docetaxel treatment only, ARM 4: Extension phase of Docetaxel arm: AEs that occurred on 3mg/kg Nivolumab, ARM 5: Extension phase of Docetaxel arm: AEs that occurred on or 480 mg Nivolumab
Groups:
- Nivolumab 3 mg/kg: Nivolumab 3 mg/kg solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
- Nivolumab 480 mg: Nivolumab 480 mg solution intravenously every 4 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
- Docetaxel: Docetaxel 75mg/m^2 solution intravenously every 3 weeks until documented disease progression , discontinuation due to toxicity, withdrawal of consent or study ends.
- Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg: Eligible patients from the Docetaxel arm may receive nivolumab 3 mg/kg every 2 weeks via extension phase until documented disease progression, discontinuation due to toxicity, withdrawal of consent or study ends.
- Extension Phase of Docetaxel Arm: Nivolumab 480 mg: Eligible patients from the Docetaxel arm may receive nivolumab 480 mg flat dose every 4 weeks via extension phase until documented disease progression, discontinuation due to toxicity, withdrawal of consent or study ends.
Arm/Group | Nivolumab 3 mg/kg | Nivolumab 480 mg | Docetaxel | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg | Extension Phase of Docetaxel Arm: Nivolumab 480 mg
All-Cause Mortality (participants affected / at risk) | 119/135 | 2/6 | 129/137 | 5/6 | 1/1
Serious Adverse Events (participants affected / at risk) | 85/131 | 1/6 | 92/129 | 4/6 | 0/1
Other Adverse Events (participants affected / at risk) | 120/131 | 4/6 | 123/129 | 4/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=131) | Nivolumab 480 mg (N=6) | Docetaxel (N=129) | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg (N=6) | Extension Phase of Docetaxel Arm: Nivolumab 480 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 13 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 4 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 14 | 1 | 17 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40 | 0 | 36 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=131) | Nivolumab 480 mg (N=6) | Docetaxel (N=129) | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg (N=6) | Extension Phase of Docetaxel Arm: Nivolumab 480 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 27 | 0 | 43 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 11 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 43 | 0 | 0
Hypothyroidism (Endocrine disorders) | 7 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 10 | 0 | 0
Constipation (Gastrointestinal disorders) | 18 | 0 | 19 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 1 | 34 | 0 | 0
Nausea (Gastrointestinal disorders) | 24 | 2 | 33 | 2 | 0
Vomiting (Gastrointestinal disorders) | 12 | 2 | 19 | 1 | 0
Asthenia (General disorders) | 25 | 1 | 27 | 1 | 0
Chest pain (General disorders) | 6 | 0 | 10 | 1 | 0
Chills (General disorders) | 9 | 1 | 2 | 1 | 0
Fatigue (General disorders) | 42 | 0 | 52 | 1 | 0
Mucosal inflammation (General disorders) | 3 | 0 | 13 | 0 | 0
Non-cardiac chest pain (General disorders) | 8 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 11 | 0 | 16 | 0 | 0
Pain (General disorders) | 8 | 1 | 6 | 0 | 0
Pyrexia (General disorders) | 27 | 0 | 26 | 3 | 0
Bronchitis (Infections and infestations) | 14 | 1 | 4 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 0 | 7 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 0 | 5 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 6 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 8 | 0 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 8 | 0 | 0
Weight decreased (Investigations) | 13 | 0 | 8 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 8 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 35 | 0 | 41 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 0 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 0 | 10 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0 | 4 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 0 | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 0 | 19 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 0 | 12 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 7 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 3 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 15 | 0 | 0
Dizziness (Nervous system disorders) | 13 | 0 | 13 | 0 | 0
Headache (Nervous system disorders) | 18 | 1 | 10 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 0 | 14 | 0 | 0
Paraesthesia (Nervous system disorders) | 5 | 0 | 9 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 0 | 7 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 1 | 24 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 | 0 | 39 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 10 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 5 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 30 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0 | 3 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 0 | 12 | 0 | 0
Hypotension (Vascular disorders) | 7 | 0 | 5 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Blepharochalasis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 4 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0
Oesophageal compression (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 1 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0 | 6 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 6 | 1 | 0
Paronychia (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 3 | 1 | 0
Blood creatinine increased (Investigations) | 6 | 0 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0 | 5 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 5 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 5 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 2 | 0 | 3 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 4 | 1 | 2 | 0 | 0
Malaise (General disorders) | 2 | 1 | 2 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.